CLINICAL TRIAL: NCT01315288
Title: A Randomized Trial of Clinical Decision Making in Asymptomatic Carotid Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACSCDM-1
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Carotid Stenosis
Keywords: Medical decision making; Asymptomatic Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Video presentation absolute risk (Active Comparator): absolute risk
  Interventions: Other: One of 6 video presentation by one of 4 presenters
- Video presentation absolute event-free survival (Active Comparator): absolute event-free survival
  Interventions: Other: One of 6 video presentation by one of 4 presenters
- Video presentation annualized absolute risk (Active Comparator): annualized absolute risk
  Interventions: Other: One of 6 video presentation by one of 4 presenters
- Video presentation relative risk (Active Comparator): relative risk
  Interventions: Other: One of 6 video presentation by one of 4 presenters
- Video presentation qualitative description (Active Comparator): qualitative description
  Interventions: Other: One of 6 video presentation by one of 4 presenters

INTERVENTIONS:
Other: One of 6 video presentation by one of 4 presenters

SUMMARY:
The purpose of this study is to determine patient variables, physician presenter variables, and information variables that might affect clinical decision making in asymptomatic carotid stenosis. The hypothesis is that information variables are the most significant determinant of clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* No known history of carotid stenosis

Exclusion Criteria:

* History of dementia
* Unable to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Decision regarding surgery | Approximately 2 minutes
  Subjects are asked to make a choice regarding surgery after watching a 30 second video.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States